CLINICAL TRIAL: NCT02515318
Title: Effects of a Physiotherapy Program in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Physiotherapy in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0056UG
Record Dates: First submitted 2015-08-01; First posted 2015-08-04 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: COPD; Exacerbation; Hospitalisation; Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Breathing Exercises; Transcutaneous Electric Nerve Stimulation; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy program (Experimental): Patients with COPD are included in this group. They will receive a physiotherapy program during the hospitalization due to acute exacerbation of COPD, additionally to the standard medical treatment
  Interventions: Other: Physiotherapy program
- Control group (Active Comparator): Patients with COPD are included in this group. They will receive the medical standard treatment during the hospitalization due to acute exacerbation of COPD.
  Interventions: Drug: Medical standard treatment

INTERVENTIONS:
Other: Physiotherapy program — The physiotherapy treatment will be performed during the hospitalization, every day during 45-60 minutes, and included: breathing exercises, electrostimulation in quadriceps with voluntary contraction and exercises with theraband.
  Other Names: Respiratory exercises; Electrostimulation
  Arms: Physiotherapy program
Drug: Medical standard treatment — The standard medical treatment consists on:
  Inhaled bronchodilators: Short acting inhaled β2 agonists ( salbutamol and terbutaline) and anticholinergic agents (ipratropium and oxitropium bromide).
  Glucocorticoids:
  Inhaled glucocorticoids including beclomethasone dipropionate, budesonide, flunisolide, fluticasone propionate and triamcinolone acetonide, depending on the expert criteria.
  - Antibiotics: The antibiotics were administered according to the GOLD criteria including the β-lactamase inhibitor and fluoroquinolones.
  Other Names: Drugs
  Arms: Control group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is projected to be the fifth leading burden of disease worldwide by the year 2020. An acute exacerbation of COPD (AECOPD) is defined as an acute event characterized by a worsening of the patient's respiratory symptoms that requires a modification in the medication. AECOPD are frequent (mean of 1-4 exacerbations each year). It increases in frequency with the severity of the disease. The objective of this study is to examine whether a physical therapy intervention can reduce impairment in patients with COPD during hospitalization due to an acute exacerbation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the leading diseases causing mortality and morbidity, despite advanced pharmacotherapy and therapeutic management.

COPD patients suffer frequent exacerbations, defined as 'acute events characterized by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medication'. Acute illness and prolonged bed rest are associated with loss of muscle mass and a significant decline in functional ability and mobility. Interventions to counteract these impairments are indicated.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis with exacerbation.
* No contraindication of physiotherapy.
* Signed written consent.
* Medical approval for inclusion

Exclusion Criteria:

* Neurological, orthopedic or heart diseases.
* Prosthetic devices in the lower limbs.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Quadriceps strength will be assessed with a portable dynamometer. The test will be performed as previously reported
Exercise capacity | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Five times sit to stand test (5STS) will be used to assess exercise capacity, 5STS is a simple assessment tool that is feasible in all healthcare settings, and may be a rapid method of assessing changes in exercise capacity in COPD and screening for poor physical functioning individuals.

SECONDARY OUTCOMES:
Respiratory function | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Spirometry is regarded as the gold standard measure of respiratory function. Spirometry will be performed according to the American Thoracic Society criteria.
Dyspnea | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Dyspnea perception will be assessed with Borg modified scale. Patients will classify their breathlessness between 0 and 10.
Health status | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  EuroQol-5D (EQ-5D) will be used to assess quality of life. EQ-5D is a generic questionnaire and consists of two parts, the EQ-5D Visual analogue scale (VAS) and the EQ-5D index. The EQ-5D VAS consists on a vertical rating scale from 0 to 100 (0 = death/worst possible health state and 100 = best possible health state). The EQ-5D index is a five-item questionnaire (mobility, self-care, usual activity, pain/discomfort and anxiety/depression). Each item has three levels: no problem, some problem and severe problem.
Fatigue | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  Fatigue will be assessed with the Fatigue Severity Scale (FSS). The FSS is a nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, querying its relationship to motivation, physical activity, work, family, and social life, and asking respondents to rate the ease with which they are fatigued and the degree to which the symptom poses a problem for them.
Impact of COPD | Participants will be followed for the duration of hospital stay, an expected average of 9 days.
  The impact of COPD in patient's life will be evaluated with COPD Assessment Test (CAT) that is a simple instrument to quantify chronic obstructive pulmonary disease (COPD) impact in routine practice.

OTHER OUTCOMES:
Dependency levels | Baseline
  Dependency levels will be evaluated with the Functional Independence Measure (FIM). It is an 18-item, 7-level scale developed to uniformly assess severity of patient disability and medical rehabilitation functional outcome.
Comorbidities | Baseline
  Charlson Comorbidity Index will be used to assess the comorbidities of the patients, it is a simple and valid method of estimating risk of death from comorbid disease. It contains 19 categories of comorbidity and predicts the ten-year mortality for a patient who may have a range of co-morbid conditions. Each condition is assigned with a score of 1, 2, 3 or 6 depending on the risk of dying associated with this condition.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - University of Granada, Granada
  - Department of Physical Therapy, Granada

IPD SHARING:
Plan to Share IPD: Undecided